CLINICAL TRIAL: NCT03423524
Title: Clinical Study to Investigate Visual Performance of a Hydrophobic Monofocal IOL After Bilateral Implantation
Acronym: PHY1801
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY1801
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Cataract; Lens Opacities
Keywords: Intraocular lens; Monofocal; Hydrophobic
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm: Investigational Device (Experimental): Implantation of monofocal intraocular lens (IOL) "Micropure 1.2.3." consisting of hydrophobic material
  Interventions: Device: Micropure 1.2.3.

INTERVENTIONS:
Device: Micropure 1.2.3. — Implantation of intraocular lens (IOL). Name: "MicroPure 1.2.3." It is a monofocal intraocular lens consisting of hydrophobic acrylic material. One IOL per eye will be implanted

SUMMARY:
Prospective, non-randomised, open, controlled, single-center post-market clinical follow study about Micropure 1.2.3 IOL.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, non-randomised, open, controlled, single-center post-market clinical follow whereby study patients undergoing routine cataract surgery will have bilateral implantation of monofocal intraocular lenses Micropure 1.2.3. (PhysIOL, Liège, Belgium)

The study purpose is to obtain clinical data on visual acuity and contrast sensitivity on patients implanted with Micropure 1.2.3.

The device under investigation (Micropure 1.2.3.) is a monofocal glistening-free hydrophobic acrylic intraocular lens (IOL) manufactured by the sponsor of this study PhysIOL sa/nv. The IOL will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

In total 50 patients will be recruited for this clinical study and receive a bilateral implantation of Micropure 1.2.3. intraocular lens.

Subjects participating in the trial will attend a total of 8 study visits (1 preoperative, 2 operative and 5 postoperative) over a period of 2 Years.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Irregular astigmatism
* Age of patient < 45 years
* Regular corneal astigmatism >0.75 dioptres by an automatic keratometer or biometer or >1.0 dioptres if the steep axis of cylinder is between 90° and 120°
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* Complicated surgery
* Patients who do not give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
monocular Corrected Distance Visual Acuity (CDVA) | 3 months postoperative
  Statistically non-inferior visual acuity outcomes on monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions compared to literature data on a monofocal hydrophilic IOL (Bausch & Lomb - Akreos MI60) at the 3 months follow up visit.

SECONDARY OUTCOMES:
Manifested refraction | 1 month, 3 months, 12 months, 24 months postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2014.
Monocular and binocular Uncorrected Distance Visual Acuity (UDVA) | 1 month, 3 months, 12 months, 24 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Monocular and binocular Uncorrected Intermediate Visual Acuity (UIVA) | 1 month, 3 months, 12 months, 24 months postoperative
  UIVA is measured with ETDRS charts placed in 70cm distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Monocular and binocular Distance Corrected Intermediate Visual Acuity (DCIVA) | 1 month, 3 months, 12 months, 24 months postoperative
  DCIVA is measured with ETDRS charts placed in 70cm distance and using best distance corrected refraction according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Binocular Corrected Distance Visual Acuity (CDVA) | 1 month, 3 months, 12 months, 24 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done binocularly
Monocular and binocular Contrast Sensitivity under photopic and mesopic light conditions | 1 month, 3 months, 12 months, 24 months postoperative
  Contrast Sensitivity under photopic and mesopic light conditions using the standardized contrast sensitivity device CSV-1000 (VectorVision)
Monocular and binocular assessment of defocus curve under photopic light conditions | 1 month, 3 months, 12 months, 24 months postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions will be measured. This test is performed with best distance corrected refraction and spherical additions ranging from -2.0 D to +1.5 D
Slitlamp examination - Corneal status | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal status.
Slitlamp examination - Fundus | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus.
Slitlamp examination - Signs of inflammation | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Signs of inflammation.
Slitlamp examination - Pupillary block | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Pupillary block.
Slitlamp examination - Retinal detachment | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Retinal detachment.
Slitlamp examination - Status of anterior and posterior capsule | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Status of anterior and posterior capsule.
Slitlamp examination - IOL decentration | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL decentration.
Slitlamp examination IOL tilt | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL tilt.
Slitlamp examination - IOL discoloration | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL discoloration.
Slitlamp examination - IOL opacity | 12 months, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL opacity.

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | Pre-operative, 1 month, 3 months, 12 months, 24 months postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations
Questionnaire on IOL implantation | peroperative
  A questionnaire will be handed out to the surgeon right after the surgery to document the ease of use and possible issues during IOL implantation. These data will be used to compare the outcomes to different surgery techniques or injectors. The questionnaire is not validated and the outcomes serve only for the sponsor to receive feedback if one or the other IOL is easier to implant.
Keratometry | preoperative
  Keratometric measurements are performed to calculate the required IOL power
Biometry | preoperative
  Biometry measurements are performed to calculate the required IOL power

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Van Cauwenberge, MD, Principal Investigator — Ophtalmology department - CHU liège
Locations (1):
- Ophtalmology department - CHU liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No